CLINICAL TRIAL: NCT00138476
Title: Evaluation of a New Challenge Pool of Norwalk Virus Inoculum (Lot 42399) in Human Subjects
Brief Title: New Challenge Pool of Norwalk Virus Inoculum
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 99-036; BCM-IRB 10690; GCRC 2027; HHSN272200800002C
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2012-04

CONDITIONS: Gastroenteritis Norovirus
Keywords: Norovirus, calicivirus, gastroenteritis, Norwalk virus, challenge
MeSH Terms: conditions — Gastroenteritis

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- Group 4: 0.48 RT-PCR units or Placebo (Experimental): Group 4: dosage group of 10 subjects will receive 0.48 RT-PCR units of Lot 42399 NV or placebo control (8 subjects will receive NV and 2 subjects will receive placebo control).
  Interventions: Drug: Placebo; Biological: Norwalk Virus
- Group 3: 4.8 RT-PCR units or Placebo (Experimental): Group 3: dosage group of 12 subjects will receive 4.8 RT-PCR units of Lot 42399 NV or placebo control (10 subjects will receive NV and 2 subjects will receive placebo control).
  Interventions: Drug: Placebo; Biological: Norwalk Virus
- Group 2: 48 RT-PCR units or Placebo (Experimental): Group 2: dosage group of 12 subjects will receive 48 RT-PCR units of Lot 42399 NV or placebo control (10 subjects will receive NV and 2 subjects will receive placebo control).
  Interventions: Drug: Placebo; Biological: Norwalk Virus
- Group 1: 4800 RT-PCR units or Placebo (Experimental): Group 1: dosage group of 11 subjects will receive 4800 reverse transcription polymerase chain reaction (RT-PCR) units of Lot 42399 Norwalk Virus (NV) or placebo control (9 subjects will receive NV and 2 subjects will receive placebo control).
  Interventions: Drug: Placebo; Biological: Norwalk Virus
- Validation Group: 4.8 and 0.48 RT-PCR units (Experimental): Validation Group: dosage group of 12 subjects, 4 will receive 4.8 RT-PCR units and 8 will receive 0.48 RT-PCR units of Lot 42399 NV. No placebo control.
  Interventions: Biological: Norwalk Virus

INTERVENTIONS:
Drug: Placebo — 120 mL of the sodium bicarbonate solution, followed by 82 mL of sterile water, United States Pharmacopeia (USP) without virus; followed by 500 mg of sodium bicarbonate aqueous solution taken 5 minutes after placebo inoculation.
  Arms: Group 1: 4800 RT-PCR units or Placebo; Group 2: 48 RT-PCR units or Placebo; Group 3: 4.8 RT-PCR units or Placebo; Group 4: 0.48 RT-PCR units or Placebo
Biological: Norwalk Virus — Prepared and packaged from liquid feces (DC544) by clarification, centrifugation, and serial dilutions; desired doses [reverse transcription polymerase chain reaction (RT-PCR) Units] 4800, 48, 4.8, 0.48.

SUMMARY:
The main objective of this study is to see the number of volunteers that get sick from a Norwalk virus (NV) inoculation with typical symptoms of nausea, vomiting, and diarrhea. If this NV preparation is shown to cause Norwalk illness, then it can be used to test new vaccines in the future. Additionally, researchers hope to determine the lowest dose of NV inoculum that can be given to volunteers and cause illness. Study participants will include 57 healthy adults, ages 18-50. Participants will either be given the NV inoculum or placebo (water without virus). Participants will be hospitalized for a maximum of 7 days and a minimum of 4 days following the NV challenge. Study procedures include physical exam, blood testing, and collection of saliva, urine, and stool samples. Participants will be involved in study related procedures for up to 180 days.

DETAILED DESCRIPTION:
Noroviruses are the cause of most acute, epidemic, non-bacterial gastroenteritis (24-hour intestinal flu) and Norwalk virus (NV) is the prototype strain of this group of viruses. Although NV was identified some 30 years ago, progress in understanding its molecular characteristics has been slow due to the inability to grow the virus in cell culture and the lack of an animal model. As such, most work must be performed in human volunteers. The principal source of virus for research has been stool samples obtained from human volunteers who were experimentally infected with NV (NIH-8fIIa) obtained from the National Institutes for Health (NIH). The quantities of NV were sufficient to characterize the entire genome and significant advances have been made. The original NV challenge pool, obtained from the NIAID/NIH, is no longer available. Using stored stool specimens obtained from an otherwise healthy subject who was infected approximately 14 years ago with NV (NIH-8fIIa), a new pool (filtrate) was produced. This study has been designed to support an IND application, for NV challenge pool Lot 42399, to be submitted by the DMID/NIAID/NIH. The safety and infectivity of the new NV challenge pool will be established by this protocol. The clinical attack rate of Lot 42399 will be determined. Initially, 20 subjects will be challenged with a dose of NV (Lot 42399) that approximates the dose used in previous challenge studies. The predicted rate of infection in this study, defined by fecal viral shedding or seroresponse, is at least 90% of those who receive inoculation. Approximately two-thirds of infected subjects are expected to become symptomatic. Subsequently, smaller groups of subjects will be challenged with lower dosages to determine the Human Infectious Dose 50 percent (HID50). The overall objective of this study is to develop a challenge pool/inoculum of NV. The specific objectives of this clinical study are: to determine the safety and acute toxicity of a new NV challenge pool; to determine the NV clinical attack rate; to determine the infection rate and HID50 of NV Lot 42399; to measure specific immunoglobulin responses to NV Lot 42399 inoculation/infection in blood, saliva and intestinal excretions; and examine peripheral blood mononuclear cells for the presence of NV. Study participants will include 57 healthy adults, ages 18-50. This double-blind study consists of informed consent, a screening and enrollment period, the NV challenge (inpatient NV inoculation phase), and a post challenge follow-up period. Many subjects participating in this study are expected to become ill with typical symptoms and signs of viral gastroenteritis. Subjects will be hospitalized, for up to a maximum of 7 days and minimum of 4 days. Participants will be involved in study related procedures for up to 180 days.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 to 50 years of age and in good health as determined by medical history and physical examination.
* Subjects must sign informed consent prior to study initiation.
* All screening clinical laboratory test results within the protocol-defined normal range. Subjects with a history of positive Hepatitis A antibody or vaccination and normal liver transaminases (serum) may be accepted.
* If the subject is a woman, a negative serum pregnancy test within 3 days of inoculation and negative urine or blood pregnancy test on day of inoculation.
* Subjects must be able to demonstrate a sufficient understanding of the study protocol and the ability to follow all required study procedures, including measures to prevent Norwalk Virus (NV) contamination of the environment and spread of NV infection and illness to the community. The prospective subjects must pass (> 75 percent correct responses, or 21 of 27 questions answered correctly) a written examination before enrollment. The exam will contain 27 multiple choice or true/false questions on all aspects of the study protocol. Subjects will be re-instructed about any question they may have answered incorrectly.
* Subjects must be available to return for follow-up visits following discharge from the General Clinical Research Center (GCRC) and deliver specimens to the investigator promptly.
* Agree to storage of unused, identifiable clinical specimens for an indefinite period at Baylor College of Medicine for use in future research.
* Subject must express the H type-1 oligosaccharide (as measured by positive salivary secretor status).
* Must use acceptable form of birth control, if female. The only acceptable birth control methods are oral contraceptives, intrauterine devices (IUDs), contraceptive implants under the skin, or contraceptive injections, and condoms with foam.

Exclusion Criteria:

* Living with or having daily contact with children age 10 years or less or a woman known to be pregnant. This includes contact at home, school, day-care, or equivalent facilities.
* Living with or having daily contact with childcare workers.
* Living with or having daily contact with elderly persons, aged 70 years or more, or the infirmed, diapered individuals, persons with disabilities or incontinent persons. This includes work or visits to nursing homes and day-care or equivalent facilities.
* Evidence of recent (within 3 months), or of current nonbacterial gastroenteritis suggestive of Norwalk Virus (NV) infection [vomiting or unformed or watery stools (>2 during a 24 hour period)].
* History of chronic functional dyspepsia, chronic gastroesophageal reflux disease, peptic ulcer disease, gastrointestinal hemorrhage, gall bladder disease, inflammatory bowel disease, irritable bowel syndrome, frequent diarrhea, or diverticulitis anytime during the subject's lifetime.
* Positive serological tests for hepatitis viruses B (core and/or surface antigen serology) and/or C, human immunodeficiency virus (HIV)-1, or syphilis. Prior to HIV-1 testing, subjects will be counseled by a qualified clinical investigator as to the purpose and meaning of such testing. Any subject with a positive test will be referred to the local HIV-1 clinic or his/her private practitioner.
* Pregnant or lactating woman.
* History of drug or alcohol dependence, or significant acute or chronic medical or psychiatric illness that could limit the subject's ability to complete the study and/or compromise the objectives of the study. One positive CAGE questionnaire response is exclusionary.
* Regular use of medication, such as, but not limited to, corticosteroids, anti-diarrhea medications, opioids, immunosuppressive agents, nonsteroidal anti-inflammatory drugs, antipyretics, and anticoagulants (e.g., warfarin or heparin or gold salts). Oral contraceptives are permitted.
* Use of antibiotics within 14 days of inoculation.
* Use of an investigational drug within 30 days prior to the start of study drug.
* Evidence of renal disease, as indicated by (any of the following) , serum sodium, or serum potassium outside normal laboratory range, or BUN or serum creatinine >upper limit of normal range, or uric acid >8.5 mg/dL.
* A baseline serum amylase value of 115 IU/L or greater or a baseline serum lipase value of 210 IU/L or greater.
* Evidence of cardiovascular disease, as indicated by (any of the following) blood pressure >150/90 mm HG in two measurements on different days, hospitalization for myocardial infarction, arrhythmia, syncope, or murmur (non-functional) detected on physical examination.
* Evidence of liver or other reticuloendothelial disease as indicated by (any of the following) serum alanine aminotransferase (ALT) > 1.25 times normal, aspartate aminotransferase (AST) > 1.25 times normal, alkaline phosphatase > 1.25 times normal, hepatosplenomegaly, jaundice, or lymphadenopathy on physical examination.
* Evidence of hematologic, rheumatologic, or immunologic disease, as indicated by (any of the following) white blood cell count <3.0 thous./cu.mm, white blood cell count >11.0 thousand/cu.mm, neutropenia (<1500/cu.mm), hemoglobin outside laboratory normal range, history of more than 3 hospitalizations for invasive bacterial infections (pneumonia, meningitis), acute or chronic dermatitis (e.g., eczema, seborrhea, psoriasis) or collagen vascular disease [e.g., systemic lupus erythematosus (SLE) or dermatomyositis].
* History or evidence of diabetes mellitus or hyperglycemia (e.g., random glucose >120 mg/dL).
* The presence of other serious chronic illness (i.e., malignancy other than a resolved skin lesion, neurological condition or malnutrition).
* Bacterial gastroenteritis or positive fecal culture for salmonella, campylobacter, E. coli 0157:H7, and Shigella; positive fecal screen for ova and parasites with fecal white cell examination.
* Employment in the food service industry, such as restaurants, or cafeteria facilities. Specifically, this will include persons whose employment requires food processing in the 4 weeks following inoculation.
* Health-care workers with patient contact expected in the 4 weeks following inoculation.
* Expected contact (through employment or at home) with immunocompromised persons (HIV-positive, receiving immunosuppressive medications such as oral steroids, anti-neoplastic agents) in the 4 weeks following inoculation.
* Employment as an airline flight attendant scheduled to work in the 4 weeks following inoculation. Persons planning on taking a cruise in the 4 weeks following inoculation.
* Persons who have consumed or plan to consume raw shellfish (e.g., oysters) within 7 days prior to enrollment or throughout the study.
* Other conditions that in the opinion of the investigator might jeopardize the safety or rights of a volunteer subject participating in the trial or would render the subject unable to comply with the study protocol.
* Expresses blood group B histoblood group antigen (blood group B or AB)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2004-08; Primary Completion 2012-04 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Determine the clinical attack rate for viral gastroenteritis induced by Norwalk Virus (NV) Lot 42399. | Up to 7 days or until clinical symptoms of diarrhea and vomiting have resolved.
Safety and acute toxicity of a new Norwalk virus challenge pool (Lot 42399) through clinical and laboratory monitoring of subjects. | Screening Days 30, 90, and 180
Determine the human infectious dose 50 percent of NV Lot 42399 based on viral shedding as measured by reverse transcription polymerase chain reaction (RT-PCR), by antigen shedding or by NV seroresponse by enzyme-linked immunosorbent assay (ELISA). | Screening, Days 2, 3, 4, 5, 6, 7, 14, 30, and 180.

SECONDARY OUTCOMES:
Measure specific IgG and IgA immunoglobulin responses to NV Lot 42399 inoculation/infection by ELISA, in serum, saliva and stool. | Screening, Days 0, 1, 2, 3, 4, 5, 6, 7, 8-13, 14, 15-21, 28, 30, 35, 42, 49, 56 and 180.
Examine peripheral blood mononuclear cells for the presence of NV genome by RT-PCR. | Screening, Days 2, 7, 14, 30 and 180.
Examine a variety of serum cytokine responses including interferon alpha, interleukin-10, C-reactive protein, TNF-alpha and IL-6 to NV infection and correlate acute, convalescent, and recovery cytokine levels with illness severity. | Screening, Days 1, 2, 3, 4, 5, 6, 7, 30, 90, and 180.
Examine stool by immune electron microscopy for NV particles. | Screening, Days 0, 1, 2, 3, 4, 5, 6, 7, 8-13, 14, 15-21, 28+/-3, 30, 35+/-3, 42+/-3, 49+/-3, and 56+/-3.

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine - Molecular Virology and Microbiology, Houston, Texas, United States

REFERENCES:
- [Result] Atmar RL, Opekun AR, Gilger MA, Estes MK, Crawford SE, Neill FH, Ramani S, Hill H, Ferreira J, Graham DY. Determination of the 50% human infectious dose for Norwalk virus. J Infect Dis. 2014 Apr 1;209(7):1016-22. doi: 10.1093/infdis/jit620. Epub 2013 Nov 18. PMID 24253285
- [Derived] Reeck A, Kavanagh O, Estes MK, Opekun AR, Gilger MA, Graham DY, Atmar RL. Serological correlate of protection against norovirus-induced gastroenteritis. J Infect Dis. 2010 Oct 15;202(8):1212-8. doi: 10.1086/656364. PMID 20815703